CLINICAL TRIAL: NCT01377480
Title: Phase 2 Proof-of-Activity Study of Oral Posaconazole in the Treatment of Asymptomatic Chronic Chagas Disease (Phase 2, Protocol No. P05267)
Brief Title: A Study of the Use of Oral Posaconazole (POS) in the Treatment of Asymptomatic Chronic Chagas Disease (P05267)
Acronym: STOP CHAGAS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P05267; MK-5592-055 (Other: Merck Protocol Number)
Record Dates: First submitted 2011-05-13; First posted 2011-06-21 (Estimated); Results first posted 2015-08-10 (Estimated); Last update posted 2018-08-27 (Actual); Status verified 2018-07

CONDITIONS: Chagas Disease
MeSH Terms: conditions — Chagas Disease | interventions — posaconazole; benzonidazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Posaconazole (Experimental): Posaconazole (POS) 400 mg (10 mL) oral suspension twice daily for 60 days
  Interventions: Drug: Posaconazole
- Placebo (Placebo Comparator): Posaconazole placebo (10 mL) oral suspension twice daily for 60 days
  Interventions: Drug: Placebo for posaconazole
- Posaconazole + Benznidazole (Experimental): Posaconazole 400 mg (10 mL) oral suspension twice daily for 60 days and benznidazole (BNZ) 100 mg oral tablet twice daily (200-mg daily dose) for 60 days
  Interventions: Drug: Posaconazole; Drug: Benznidazole
- Benznidazole + Placebo (Active Comparator): Posaconazole placebo (10 mL) oral suspension twice daily for 60 days and benznidazole 100 mg oral tablet twice daily (200-mg daily dose) for 60 days
  Interventions: Drug: Placebo for posaconazole; Drug: Benznidazole

INTERVENTIONS:
Drug: Posaconazole — POS 40 mg/mL oral suspension
  Other Names: SCH 056592, MK-5592
  Arms: Posaconazole; Posaconazole + Benznidazole
Drug: Placebo for posaconazole — Placebo oral suspension
  Arms: Benznidazole + Placebo; Placebo
Drug: Benznidazole — BNZ 100 mg oral tablet
  Arms: Benznidazole + Placebo; Posaconazole + Benznidazole

SUMMARY:
This is a study to compare the efficacy of oral posaconazole to placebo for the treatment of asymptomatic Chagas disease. The primary hypothesis of the study is that posaconazole 400 mg twice daily improves therapeutic response compared to placebo in participants with a diagnosis of asymptomatic chronic Chagas disease.

ELIGIBILITY:
Inclusion Criteria:

- Must have a positive serology result for Trypanosoma cruzi on any 2 of 3 of the following tests: indirect immunofluorescence, indirect hemagglutination, or enzyme-linked immunoabsorbent assay (ELISA)

* Must have a positive qualitative polymerase chain reaction (PCR) for Trypanosoma cruzi
* Must have a normal 12-lead electrocardiogram (ECG)
* Must have a normal 2-D echocardiogram
* Must have no evidence of ventricular tachycardia on 24-hour Holter monitoring
* Female participants of childbearing age must be using a medically accepted method of birth control before beginning study drug treatment and must agree to continue its use during the study, or must have been surgically sterilized
* Female participants of childbearing potential must have a negative serum beta-human chorionic gonadotropin (hCG) pregnancy test at Screening and a negative urine pregnancy test at Baseline or within 72 hours before the start of study drug

Exclusion Criteria:

* Are breastfeeding, pregnant, or planning to become pregnant
* Body weight <60 kg
* Have an immunodeficiency or are immunosuppressed
* History of megacolon with obstipation or megaesophagus with severe swallowing impairment.
* Have previously received treatment with benznidazole or nifurtimox
* Known allergy/sensitivity to azoles
* Has aspartate aminotransferase (AST) or alanine aminotransferase (ALT) levels greater than 2.5 times the upper limit of normal at Screening
* Has serum creatinine >2.5 mg/dL or 200 micromoles at Screening
* Has a history of severe alcohol abuse within two years from Screening
* Is taking any of the prohibited medication

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2011-07-06 (Actual); Primary Completion 2014-07-22 (Actual); Study Completion 2015-01-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Morillo CA, Waskin H, Sosa-Estani S, Del Carmen Bangher M, Cuneo C, Milesi R, Mallagray M, Apt W, Beloscar J, Gascon J, Molina I, Echeverria LE, Colombo H, Perez-Molina JA, Wyss F, Meeks B, Bonilla LR, Gao P, Wei B, McCarthy M, Yusuf S; STOP-CHAGAS Investigators. Benznidazole and Posaconazole in Eliminating Parasites in Asymptomatic T. Cruzi Carriers: The STOP-CHAGAS Trial. J Am Coll Cardiol. 2017 Feb 28;69(8):939-947. doi: 10.1016/j.jacc.2016.12.023. PMID 28231946
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=P05267&kw=P05267&tab=access

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 393 participants were screened, 123 were eligible for enrollment, and 120 were randomized
Groups:
- Posaconazole: POS 400 mg (10 mL) oral suspension twice daily for 60 days
- Placebo: POS placebo (10 mL) oral suspension twice daily for 60 days
- Posaconazole + Benznidazole: POS 400 mg (10 mL) oral suspension twice daily for 60 days and BNZ 100 mg oral tablet twice daily (200-mg daily dose) for 60 days
- Benznidazole + Placebo: BNZ 100 mg oral tablet twice daily (200-mg daily dose) for 60 days and POS placebo (10 mL) oral suspension twice daily for 60 days
Period: Overall Study
Arm/Group | Posaconazole | Placebo | Posaconazole + Benznidazole | Benznidazole + Placebo
Started | 32 (Includes 2 participants randomized to POS + BNZ but who only received POS) | 30 | 28 (2 participants received only POS and were analyzed as part of the posaconazole group) | 30
Completed | 32 | 29 | 18 | 19
Not Completed | 0 | 1 | 10 | 11
Not completed — Protocol Violation | 0 | 0 | 0 | 4
Not completed — Evidence of drug-induced hepatotoxicity | 0 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0
Not completed — Serious adverse event | 0 | 0 | 1 | 1
Not completed — Other | 0 | 0 | 7 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Posaconazole | Placebo | Posaconazole + Benznidazole | Benznidazole + Placebo | Total
Number analyzed (Participants) | 32 | 30 | 28 | 30 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.3 (8.6) | 42.2 (7.8) | 40.2 (8.4) | 40.4 (7.7) | 40.8 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 7 | 13 | 17 | 53
  Male | 16 | 23 | 15 | 13 | 67

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Successful Response as Measured by Qualitative Polymerase Chain Reaction
Description: Blood samples were collected for qualitative polymerase chain reaction (PCR) assay for Trypanosoma cruzi deoxyribonucleic acid (DNA). Successful response was defined as a negative qualitative PCR value at the Day 180 follow up visit.
Time Frame: Day 180
Population: The Full Analysis Population included all randomized subjects who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Posaconazole | Placebo | Posaconazole + Benznidazole | Benznidazole + Placebo
Number analyzed (Participants) | 32 | 30 | 28 | 30
Percentage of participants | 15.6 [6.9 to 31.8] | 10.0 [3.5 to 25.6] | 82.1 [64.4 to 92.1] | 86.7 [70.3 to 94.7]

ADVERSE EVENTS:
Time Frame: All adverse events: up to Day 90 (30 days post treatment); procedure-related serious adverse events: up to Day 360 (300 days post treatment)
Arm/Group | Posaconazole | Placebo | Posaconazole + Benznidazole | Benznidazole + Placebo
Serious Adverse Events (participants affected / at risk) | 1/32 | 1/30 | 2/28 | 3/30
Other Adverse Events (participants affected / at risk) | 12/32 | 8/30 | 18/28 | 21/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Posaconazole (N=32) | Placebo (N=30) | Posaconazole + Benznidazole (N=28) | Benznidazole + Placebo (N=30)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Photodermatosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Posaconazole (N=32) | Placebo (N=30) | Posaconazole + Benznidazole (N=28) | Benznidazole + Placebo (N=30)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 1 (1) | 5 (7) | 3 (4)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (3) | 2 (3)
Asthenia (General disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Nasopharyngitis (Infections and infestations) | 2 (2) | 1 (1) | 3 (3) | 0 (0)
Transaminase increased (Investigations) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 3 (3) | 2 (2)
Headache (Nervous system disorders) | 3 (4) | 2 (3) | 8 (14) | 4 (5)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 4 (5) | 6 (8)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees to provide to the sponsor 45 days prior to submission for publication or presentation, review copies of abstracts or manuscripts for publication that report any results of the trial. The sponsor shall have the right to review and comment with respect to publications, abstracts, slides, and manuscripts with regard to proprietary information, accuracy, and fair-balance and compliance.